CLINICAL TRIAL: NCT07055139
Title: Comparison of Digital Versus Traditional Aftercare for Uncomplicated Distal Radius and Clavicle Fractures
Brief Title: Digital Aftercare for Wrist and Clavicle Fractures
Acronym: DA-DRAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00830
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Distal Radius Fracture; Clavicle Fracture; Postoperative Care; Patient-Reported Outcome Measures (PROMs); Upper Extremity Fractures
Keywords: distal radius fracture; clavicle fracture; digital aftercare; app-based aftercare; App-Based Rehabilitation; Wrist Fracture; Fracture Recovery; Functional Outcome; QuickDASH; PRWE; eHealth; Patient Satisfaction; Quality of Life; EQ-5D; Complication Rate; Postoperative Care
MeSH Terms: conditions — Wrist Fractures; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Aftercare (Active Comparator): Participants receive standard postoperative follow-up care, including scheduled clinical visits and in-person physiotherapy sessions, in accordance with institutional guidelines. Rehabilitation is delivered face-to-face and tailored to fracture type and recovery progress.
  Interventions: Behavioral: Traditional Aftercare
- Digital Aftercare (Experimental): A digital follow-up protocol delivered through a mobile app, focusing on independent functional recovery with physiotherapy exercises, educational modules, and symptom monitoring. Participants are guided through a week-by-week recovery plan specific to the fracture type.
  Interventions: Behavioral: Digital Aftercare

INTERVENTIONS:
Behavioral: Digital Aftercare — A structured, app-based digital aftercare program designed for patients recovering from distal radius or clavicle fractures. The 12-week program includes weekly video-guided physiotherapy exercises, educational content on fracture healing, pain management guidance, and milestone-based progression. The program replaces in-person physiotherapy and standard clinic follow-up, with patients instructed to follow the app independently. Medical contact is initiated only in case of uncertainty or complications.
  Arms: Digital Aftercare
Behavioral: Traditional Aftercare — Standard postoperative follow-up care for patients with distal radius or clavicle fractures, consisting of scheduled clinical visits and in-person physiotherapy sessions according to institutional protocols. The treatment includes individual exercise instruction, physiotherapy, and physician-led follow-up at defined intervals during the 12-week rehabilitation period.
  Arms: Traditional Aftercare

SUMMARY:
This prospective, two-arm, open-label clinical trial compares digital aftercare with traditional follow-up in adult patients after surgical treatment of uncomplicated distal radius or clavicle fractures. The primary objective is to assess functional recovery at three months, using the Patient-Rated Wrist Evaluation (PRWE) for wrist fractures and the QuickDASH for clavicle fractures. Secondary outcomes include range of motion, patient satisfaction, quality of life, complication rates, healthcare costs, and work disability. In the digital aftercare group, program adherence and user experience will also be evaluated through app usage data and a structured questionnaire. The study aims to determine whether digital aftercare is a clinically and economically equivalent alternative to standard in-person care.

DETAILED DESCRIPTION:
This is a prospective, open-label, two-arm clinical trial designed to compare digital aftercare with traditional in-person follow-up in adult patients (aged 18-65) who have undergone uncomplicated surgical treatment for distal radius or clavicle fractures.

Participants in the digital aftercare group receive a structured, app-based rehabilitation program over 12 weeks. The program includes video-guided physiotherapy exercises, educational content, and recovery milestones. Clinical follow-up and physiotherapy are replaced by the digital program, with medical consultations available only if clinically necessary. Adherence and user experience are tracked via app usage data and a structured questionnaire.

Participants in the traditional aftercare group receive standard postoperative care, including regular clinical follow-up visits and supervised physiotherapy sessions based on institutional guidelines.

The primary objective of this study is to evaluate whether digital aftercare results in equivalent functional outcomes compared to traditional follow-up. Functional recovery is assessed at 12 weeks using the QuickDASH (for clavicle fractures) and PRWE (for distal radius fractures).

Secondary outcomes include range of motion, patient satisfaction (VAS), quality of life (EQ-5D), complication rates (Clavien-Dindo classification), direct and indirect healthcare costs, return to work, and - in the digital group - program adherence and user feedback.

This study also aims to explore the cost-effectiveness of digital aftercare and its potential as a scalable alternative to traditional rehabilitation in selected fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Surgically treated, uncomplicated distal radius or clavicle fracture
* Use of a smartphone (iOS or Android)
* Ability to understand German and complete study-related questionnaires
* Provided written informed consent

Exclusion Criteria:

* Polytrauma or additional injuries to the same upper extremity
* No access to or inability to use a smartphone
* Cognitive, psychiatric, or language barriers impairing participation
* Pregnancy
* Inability or unwillingness to comply with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional Recovery at 12 Weeks (PRWE for distal radius) | 12 weeks postoperatively
  Functional outcome will be assessed using the Patient-Rated Wrist Evaluation (PRWE) score. The PRWE is a validated questionnaire specifically designed to evaluate wrist function and pain. Scores range from 0 to 100, with lower scores indicating better functional outcomes.
Functional Recovery at 12 Weeks (QuickDASH for clavicle) | 12 weeks postoperatively
  Functional outcome will be assessed using the QuickDASH (Disabilities of the Arm, Shoulder and Hand - Short Version) score. The QuickDASH is a validated tool to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. Scores range from 0 to 100, with lower scores indicating better function.

SECONDARY OUTCOMES:
Range of Motion | 12 weeks postoperatively
  Goniometric assessment of wrist or shoulder range of motion in degrees, depending on fracture type.
Patient Satisfaction | 12 weeks postoperatively
  Patient satisfaction measured using a Visual Analogue Scale (VAS, 0-10), with higher scores indicating greater satisfaction.
Health-Related Quality of Life | 12 weeks postoperatively
  Health-related quality of life will be measured using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. The EQ-5D-5L assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Index scores typically range from less than 0 (where 0 represents a health state equivalent to death and negative values represent health states worse than death) to 1 (representing full health). Higher scores indicate better health-related quality of life.
Complication Rates | 12 weeks postoperatively
  Surgical and postoperative complications classified according to the Clavien-Dindo classification system.
Healthcare Costs | 12 weeks postoperatively
  Direct and indirect healthcare costs associated with each aftercare modality, including physiotherapy, consultations, and work absence.
Work Disability | 12 weeks postoperatively
  Duration of work absence stratified by job type (manual vs. non-manual work).
User Experience with Digital Program (Digital Group Only) | 12 weeks postoperatively
  Assessed with a structured questionnaire on usability, satisfaction, and perceived helpfulness of the app-based program.
Number of Completed Exercise Sessions in Digital Program (Digital Group Only) | 12 weeks postoperatively
  Adherence to the digital rehabilitation program will be measured by the number of completed exercise sessions recorded via the app. One session is counted as completed when all scheduled exercises for a given day are marked as done by the user.
Login Frequency in Digital Program (Digital Group Only) | 12 weeks postoperatively
  App usage will be monitored by tracking the total number of logins to the digital rehabilitation platform over the 12-week period. Each login is defined as a unique user access within a 24-hour window.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Beeres, Prof. MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland